CLINICAL TRIAL: NCT01039194
Title: A Study of the Effect of Concomitant Administration of Multiple Doses of BMS-708163 on the Pharmacokinetics of Galantamine in Healthy Subjects
Brief Title: Drug-Drug Interaction to Study the Effect of BMS-708163 on Pharmacokinetics (PK) of Galantamine Extended Release (ER)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CN156-009
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Galantamine; BMS 708163

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- galantamine 8 mg (ER) (Active Comparator)
  Interventions: Drug: galantamine
- galantamine 16 mg (ER) (Active Comparator)
  Interventions: Drug: galantamine
- BMS-708163 (Active Comparator)
  Interventions: Drug: BMS-708163

INTERVENTIONS:
Drug: galantamine — Capsule, Oral, 8 mg (ER), once daily, Days 1-7
  Other Names: Razadyne ER ™
  Arms: galantamine 8 mg (ER)
Drug: galantamine — Capsule, Oral, 16 mg (ER), once daily, Days 8-24
  Other Names: Razadyne ER ™
  Arms: galantamine 16 mg (ER)
Drug: BMS-708163 — Capsule, Oral, 125 mg, once daily, Days 15-24
  Arms: BMS-708163

SUMMARY:
The purpose of the study is to find out if the plasma concentration of galantamine extended release is changed when BMS-708163 is administered at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and postmenopausal women

Exclusion Criteria:

* Gastrointestinal disorders
* Bleeding disorders
* Peptic ulcer disease
* Cholecystectomy
* Seizure disorder
* Asthma
* Chronic obstructive pulmonary disease
* Urinary tract obstruction
* Cardiac conduction abnormalities, including but not limited to "sick sinus syndrome" and those with unexplained syncopal episodes
* Inability to tolerate oral medication
* Inability to be venipunctured and/or tolerate venous access

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Galantamine alone and with BMS-708163: Galantamine PK parameters (Cmax, Tmax, AUC(TAU) and Ctrough rations will be assessed without BMS-708163 Day 14) and with BMS708-163 (Ctrough Day 24) | Study Days 14 & 24

SECONDARY OUTCOMES:
Galantamine alone and with BMS 708163: Safety and tolerability (AE's, ECG, vital signs, safety labs) | Study Days 7, 14, 18, 25 and study discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Parexel International - Baltimore Epcu, Baltimore, Maryland, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx